CLINICAL TRIAL: NCT05749887
Title: Salvage Surgery for Patients With Residual Disease After Concurrent Chemoradiation Therapy for Locally Advanced Cervical Cancer: A Prospective, Single-arm Clinical Study.
Brief Title: The Efficacy of Salvage Surgery in Patients With Residual Tumor After Concurrent Chemoradiation for Locally Advanced Cervical Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0112
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer
Keywords: Locally advanced cervical cancer; chemoradiotherapy; redsidual tumor; salvage sugery; OS
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- salvage sugery (Other): Salvage surgery for patients diagnosed locally advanced cervical cancr with residual tumor after standard chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy+ brachytherapy)
  Interventions: Procedure: salvage surgery

INTERVENTIONS:
Procedure: salvage surgery — Open/minimally invasive salvage surgery performed when cervical biopsy and/or PET/CT scan ( SUVmax ≥2.5 ) indicate patients with residual tumor intrapelvic 4-12 weeks after standard CCRT.
  Surgery type:
  1. No parametrial involvement, extrafascial hysterectomy;
  2. There is parametrial involvement, extensive hysterectomy(Q-MC);
  3. Only bladder invasion, anterior pelvic exenteration;
  4. Only rectal invasion, posterior pelvic exenteration or total pelvic exenteration;
  5. Invasion of bladder and rectum, total exenteration.
  6. The pelvic lymph nodes are removed at the same time when 18F -FDG PET /CT indicates that the SUVmax is ≥ 2.5.

SUMMARY:
This is a single-center single-arm study. The main purpose of this study is to study the efficacy of surgical treatment for patients with locally advanced cervical cancer (FIGO IB3, IIA2-IVA) who still have residual tumor after concurrent radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Stage Ib3 and IIA2-IVA (FIGO2018) cervical cancer with histopathology of squamous cell carcinoma, adenosquamous cell carcinoma, adenocarcinoma.
2. Complete standard CCRT(Pelvic EBRT+ concurrent platinum-containing chemotherapy+ brachytherapy).
3. After 4-12 weeks of treatment, the cervical biopsy pathology confirmed residual cancer, or the cervical biopsy was negative, but PET /CT showed that SUVmax of the residual lesions in the cervical and/or pelvic lymph nodes were ≥ 2.5, two or more gynaecological oncologists with Grade IV operation qualification and the title of deputy director or above have gynecological examination, and the multidisciplinary team(MDT) evaluation recommended surgical treatment.
4. ECOG score:0 ~ 1.
5. The expected survival time>6 months;
6. There is no absolute contraindication of surgery and the patients with good compliance.

Exclusion Criteria:

1. The radiotherapy and chemotherapy are not completed or the radiotherapy dose is not reached.
2. PET /CT and/or pathological indicates that there is a distant metastasis including para-aortic lymph nodes.
3. Other malignancies were diagnosed within five years or needed treatments.
4. History of important organ transplantation.
5. History of immune disease who need to take immunosuppressive drugs.
6. History of serious mental illness and brain functional disorder.
7. Drug abuse or drug use history.
8. Participants in other clinical trials at the same time.
9. Those who are unable or unwilling to accept surgical treatment/sign informed consent/comply with research requirements.
10. Without surgical conditions: 1) Chronic renal insufficiency or renal failure; 2) Liver insufficiency; 3)Chronic lung disease with restrictive respiratory dysfunction; 4) Cardiac dysfunction (patients with relative and absolute contraindications to surgery after consultation by cardiac physicians.
11. Patients who cannot understand the research regimen and refuse to sign the informed consent form.
12. Other concomitant diseases or special conditions seriously endanger the patient's health or interfere with the trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | 5 years
  5 years overall survival

SECONDARY OUTCOMES:
PFS | 2 years
  Progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, PH.D, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China